CLINICAL TRIAL: NCT00098423
Title: A Phase I And Pharmacological Trial Of 17-Allylamino -17-demethoxygeldanamycin (17-AAG) And Cytarabine In Refractory Leukemia And Myelodysplastic Syndrome
Brief Title: Tanespimycin and Cytarabine in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia, Acute Lymphoblastic Leukemia, Chronic Myelogenous Leukemia, Chronic Myelomonocytic Leukemia, or Myelodysplastic Syndromes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00056; NCI-2009-00056 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-6383; CDR0000401509; MC0313 (Other: Mayo Clinic); 6383 (Other: CTEP); U01CA070095 (NIH); U01CA069912 (NIH); NCT01646931 (obsolete NCT alias); NCT01664338 (obsolete NCT alias)
Record Dates: First submitted 2004-12-07; First posted 2004-12-08 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia; Adult Acute Basophilic Leukemia; Adult Acute Eosinophilic Leukemia; Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Blastic Phase Chronic Myelogenous Leukemia; Chronic Myelomonocytic Leukemia; de Novo Myelodysplastic Syndromes; Previously Treated Myelodysplastic Syndromes; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Refractory Anemia With Excess Blasts in Transformation; Relapsing Chronic Myelogenous Leukemia; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Leukemia, Basophilic, Acute; Leukemia, Eosinophilic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute; Blast Crisis; Leukemia, Myelomonocytic, Chronic; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — tanespimycin; Cytarabine

ARMS (1):
- Treatment (chemotherapy) (Experimental): Patients receive induction therapy comprising cytarabine IV continuously on days 1-5 and tanespimycin IV over 1 hour on days 3 and 6.
  Patients achieving a morphologic complete response with CRi or partial response may be eligible to receive a second induction course of therapy after day 21 at the discretion of the principal investigator. Patients achieving a CR receive up to 4 courses of consolidation therapy with cytarabine and tanespimycin. Consolidation therapy repeats approximately every 60 days in the absence of disease progression or unacceptable toxicity. Patients who achieve CR and remain in remission for â¥ 6 months may be retreated with cytarabine and tanespimycin (at the current dose level or the MTD) at the time of relapse. Cohorts of 3-6 patients receive escalating doses of tanespimycin until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Patients are followed at 3 months.
  Interventions: Drug: tanespimycin; Drug: cytarabine

INTERVENTIONS:
Drug: tanespimycin — Given IV
  Other Names: 17-AAG
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside

SUMMARY:
This phase I trial is studying the side effects and best dose of tanespimycin when given with cytarabine in treating patients with relapsed or refractory acute myeloid leukemia, acute lymphoblastic leukemia, chronic myelogenous leukemia, chronic myelomonocytic leukemia, or myelodysplastic syndromes. Drugs used in chemotherapy, such as tanespimycin and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Tanespimycin may also help cytarabine kill more cancer cells by making cancer cells more sensitive to the drug. Giving tanespimycin together with cytarabine may kill more cancer cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose of 17-N-allylamino-17-demethoxygeldanamycin (17-AAG) (tanespimycin) when administered with cytarabine in patients with relapsed or refractory acute myeloid leukemia, acute lymphoblastic leukemia, chronic myelogenous leukemia, chronic myelomonocytic leukemia, or high-grade myelodysplastic syndromes.

II. Determine the toxic effects of this regimen in these patients. III. Determine, preliminarily, the activity of this regimen in these patients. IV. Correlate the pharmacokinetics of this regimen with cytochrome p450 3A5 genotype in these patients.

V. Determine the effect of this regimen on client proteins in vivo and ex vivo using leukemic blasts from patients treated with this regimen.

OUTLINE: This is a multicenter, dose-escalation study of tanespimycin.

Patients receive induction therapy comprising cytarabine intravenously (IV) continuously on days 1-5 and tanespimycin IV over 1 hour on days 3 and 6.

Patients achieving a morphologic complete response with incomplete blood count recovery (CRi) or partial response may be eligible to receive a second induction course of therapy after day 21 at the discretion of the principal investigator. Patients achieving a complete response (CR) receive up to 4 courses of consolidation therapy with cytarabine and tanespimycin. Consolidation therapy repeats approximately every 60 days in the absence of disease progression or unacceptable toxicity. Patients who achieve CR and remain in remission for ≥ 6 months may be retreated with cytarabine and tanespimycin (at the current dose level or the maximum tolerated dose [MTD]) at the time of relapse. Cohorts of 3-6 patients receive escalating doses of tanespimycin until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Patients are followed at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of 1 of the following:

  * Acute myeloid leukemia, except acute promyelocytic leukemia (M3 disease), meeting 1 of the following criteria:

    * Failed to achieve complete remission (CR) after initial induction therapy regimen*
    * First relapse within 1 year of initial CR
    * Failed re-induction therapy at first or second relapse
    * Second or third relapse after completing ≤ 3 different induction therapy regimens
    * Antecedent hematologic disorder (myelodysplastic syndromes [MDS], chronic myeloproliferative disease, or chronic myelomonocytic leukemia [CMML])
    * Received prior chemotherapy for a non-hematologic malignancy
    * High-risk cytogenetic abnormalities (abnormalities of chromosome 5, 7, 8, or 11 OR ≥ 3 karyotypic abnormalities)
  * Acute lymphoblastic leukemia, meeting 1 of the following criteria:

    * Failed to achieve CR after initial induction therapy regimen
    * First relapse within 1 year of initial CR
    * Failed re-induction therapy at first or second relapse
    * Second or third relapse after completing ≤ 3 different induction therapy regimens
  * Chronic myelogenous leukemia, meeting the following criteria:

    * Accelerated OR blast phase (> 10% increase in the blast percentage in bone marrow)
    * Failed prior imatinib mesylate

      * No more than 1 prior chemotherapy regimen in addition to imatinib mesylate
  * CMML, meeting the following criteria:

    * More than 10% increase in blast percentage AND organ infiltration OR impending marrow failure as evidenced by cytopenia
    * No t(5;12) by cytogenetics (unless failed prior trial of imatinib mesylate)
  * High-grade MDS, defined as > 10% blasts on marrow cellularity (refractory anemia with excess blasts in transformation) OR International Prognostic Scoring System MDS prognostic score > 1.5
* Not a candidate for allogenic bone marrow transplantation* from a related sibling donor (i.e., HLA-identical sibling)
* No known standard or potentially curative therapy exists or is capable of extending life expectancy
* No clinical symptoms suggesting CNS leukemia
* Performance status - ECOG 0-2
* At least 60 days
* See Disease Characteristics
* Bilirubin ≤ 1.5 times upper limit of normal (unless attributed to underlying disease)
* Creatinine clearance ≥ 60 mL/min
* No New York Heart Association class III-IV heart failure
* No myocardial infarction within the past year
* LVEF ≥ 40% by MUGA
* No cardiac symptoms ≥ grade 2
* No uncontrolled dysrhythmia requiring medication
* No poorly controlled angina
* QTc ≤ 450 msec for men and ≤ 470 msec for women
* No congenital long QT syndrome
* No left bundle branch block
* No ischemic heart disease within the past 6 months
* No history of cardiac toxicity after treatment with anthracyclines (e.g., doxorubicin hydrochloride, daunorubicin hydrochloride, mitoxantrone hydrochloride, bleomycin, or carmustine
* No other significant cardiac disease
* No active uncontrolled infection
* No history of serious allergic reaction to eggs
* No known HIV infection or AIDS (with or without highly active antiretroviral treatment)
* DLCO > 80%
* No pulmonary symptoms ≥ grade 2
* No symptomatic pulmonary disease requiring medication including any of the following:

  * Dyspnea on or off exertion
  * Paroxysmal nocturnal dyspnea
  * Significant pulmonary disease (e.g., chronic obstruction/restrictive pulmonary disease)
* No oxygen requirement

  * No home oxygen that meets the medicare requirement
* No history of pulmonary toxicity after treatment with anthracyclines (e.g., doxorubicin hydrochloride, daunorubicin hydrochloride, mitoxantrone hydrochloride, bleomycin, or carmustine
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No psychosis
* No other serious underlying medical condition that would preclude study participation
* No prior allogeneic or autologous bone marrow transplantation
* No concurrent immunotherapy
* No concurrent biologic agents
* No concurrent gene therapy
* See Disease Characteristics
* Recovered from prior chemotherapy
* At least 48 hours since prior hydroxyurea for prevention of leukostasis
* No other concurrent chemotherapy
* At least 48 hours since prior glucocorticoids for prevention of leukostasis
* No prior radiotherapy that included the heart in the field (e.g., mantle) or chest
* No concurrent radiotherapy
* No concurrent drugs that may cause QTc prolongation
* No concurrent participation in another clinical trial involving a pharmacologic agent for symptom control or therapeutic intent
* No other concurrent investigational drugs or therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2004-11; Primary Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Tolerability of tanespimycin with cytarabine in patients with relapsed or refractory acute myeloid leukemia, acute lymphoblastic leukemia, chronic myelogenous leukemia, chronic myelomonocytic leukemia, or high-grade myelodysplastic syndromes | Day 21
  Evaluated using the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 standard toxicity grading.

SECONDARY OUTCOMES:
Clinical response | Every 2 weeks
  Evaluated as suggested by the International Working Group for Diagnosis, Standardization of Response Criteria, Treatment Outcomes and Reporting Standards for Therapeutic Trials in Acute Myeloid Leukemia. Summarized by simple descriptive summary statistics across all patients in each group as well as by dose level. Possible relationships between response and dose level will be explored graphically.
Plasma level of tanespimycin | Day 3
  Summarized by simple descriptive summary statistics across all patients in each group as well as by dose level. Possible relationships between pharmacokinetic (PK) parameters and p450 3A5 genotypes will be explored.
Effects on client proteins | Days 1, 3, and 4 of course 1
  Analyzed by immunoblotting. Results will be displayed graphically and analyzed using simple descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Kaufmann, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Kaufmann SH, Karp JE, Litzow MR, Mesa RA, Hogan W, Steensma DP, Flatten KS, Loegering DA, Schneider PA, Peterson KL, Maurer MJ, Smith BD, Greer J, Chen Y, Reid JM, Ivy SP, Ames MM, Adjei AA, Erlichman C, Karnitz LM. Phase I and pharmacological study of cytarabine and tanespimycin in relapsed and refractory acute leukemia. Haematologica. 2011 Nov;96(11):1619-26. doi: 10.3324/haematol.2011.049551. Epub 2011 Jul 26. PMID 21791475